CLINICAL TRIAL: NCT06230042
Title: Parylene-Coated Versus Silicone Catheters in the Prevention of Urinary Tract Infections and Crystallization: A Single-Center Randomized Controlled Trial
Brief Title: Catheter in the Prevention of Urinary Tract Infections and Crystallization Study(CPUTICS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CPUTICS-01
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Urinary Catheter
Keywords: urinary tract infections; urinary tract crystallization
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, the investigator and the outcomes assessor were all masked. Only the care provider who performed the anaesthesia were not blinded but they were not involved in the subsequent prostate biopsy, pain assessment, data collection and data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parylene-Coated Catheter (Experimental): The type of catheter used during a patient's indwelling urinary catheterization is Parylene-Coated Catheter
  Interventions: Other: Types of catheters
- Silicone Catheter (Active Comparator): The type of catheter used during a patient's indwelling urinary catheterization is Silicone Catheter
  Interventions: Other: Types of catheters

INTERVENTIONS:
Other: Types of catheters — One type of catheters were used for patients

SUMMARY:
This is a single-center randomized controlled trial in comparison of Parylene-Coated versus Silicone Catheters in the Prevention of Urinary Tract Infections and Crystallization.

DETAILED DESCRIPTION:
This study was a single-center randomized controlled trial, enrolling patients with indwelling urinary catheterization time greater than 2 weeks, and comparing the incidence of urinary tract infections in the two groups with different indwelling urinary catheter times by retaining mid-stream urine specimens for bacterial cultures on the 3rd, 7th, 10th, and 14th days after urinary catheter placement. And after removal of the urinary catheter,1-cm sections were taken from the head end and center of each urinary catheter, and the crystal deposition inside the catheter was observed using a scanning electron microscope. The incidence of urinary tract infections and crystal deposition on the inner wall of the catheter were compared between the patients in the matte catheter group (Parylene-coated) and the patients in the glossy catheter group (plain silicone) during the period of catheterization, so as to evaluate the effectiveness of the two types of catheters in the clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. age greater than 18 years;
2. indwelling urinary catheter for ≥14 days;
3. fully understand the clinical trial protocol and sign the informed consent;

Exclusion Criteria:

1. patients with confirmed urinary tract infection before indwelling urinary catheter;
2. those with renal dysfunction;
3. those who are allergic to silicone or silicone material;
4. those with low immunity susceptible to infection;
5. those who have participated in other clinical trials within 3 months;
6. others who are judged by the investigator to be unsuitable for clinical trials;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Catheter-Associated Urinary Tract Infection (CAUTI) Incidence | the Day 3,Day 7, Day 10 and Day 14 after catheterization
  The mid-stream urine specimens on the 3rd, 7th, 10th and 14th days after catheterization were taken for bacterial culture to compare the incidence of urinary tract infections in the two groups at different times of indwelling urinary catheterization.
  Diagnostic criteria: patients with urinary tract infections that occurred after indwelling urinary catheterization, or within 48 h of catheter removal. Urine bacterial culture of Gram-positive cocci colonies ≥104cfu/ml and Gram-negative bacilli colonies ≥105cfu/ml was judged as urinary tract infection.
Crystal deposits on the inner wall of the catheter | Day 14 after catheterization
  ① After removing the urinary catheter, a 1-cm section was taken from the head end and the center of each urinary catheter, and the crystal deposition inside the catheter was observed using a scanning electron microscope, and the average scores of the two groups were calculated according to the scores in the table below, comparing the effectiveness of the two groups of urinary catheters in preventing crystallization. ② Record the details and number of blockages that occurred during the indwelling catheterization period, and calculate the blockage rate of the two groups.

SECONDARY OUTCOMES:
Evaluation of urethral irritation response | Day 1 after catheterization
  Patients were asked about their feelings after 24h of indwelling catheterization, and the occurrence of urethral irritation reaction was recorded according to their subjective feelings.
Measuring the temperature of bladder urine | the Day 3,Day 7, Day 10 and Day 14 after catheterization
  The temperature of bladder urine was detected and recorded by connecting the machine end of the temperature measuring probe to the corresponding interface of the monitor on the 3rd, 7th, 10th, and 14th days after the patient's indwelling urinary catheter.

CONTACTS AND LOCATIONS:
Overall Officials: haifeng wang, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Once available, the results of this trial will be disseminated to an international peer-reviewed journal and presentations at international or national academic conferences. The data will be made available upon request to researchers a) who provide a methodologically sound proposal and b) whose proposed use of the data has been approved by an independent ethical review committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after publication with no end date